CLINICAL TRIAL: NCT02456025
Title: Topical Tacrolimus in Vernal Keratoconjunctivitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Eye Center and The Eye Foundation for Research in Ophthalmology (Other)
Responsible Party: Principal Investigator, Samir S. Shoughy, MD, FRCS (Glasg.), Ophthalmologist, The Eye Center and The Eye Foundation for Research in Ophthalmology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TEC 124
Record Dates: First submitted 2013-08-18; First posted 2015-05-28 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Vernal Keratoconjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical tacrolimus (Active Comparator): 20 eyes with active Vernal Keratoconjunctivitis
  Interventions: Drug: Topical tacrolimus
- Placebo (Placebo Comparator): 20 eyes with active Vernal Keratoconjunctivitis
  Interventions: Drug: Topical tacrolimus

INTERVENTIONS:
Drug: Topical tacrolimus — Topical tacrolimus 0.01% twice daily for one month
  Other Names: Tacrolimus eye drops

SUMMARY:
The main aim of this study is to evaluate the efficacy and safety of topical tacrolimus 0.01% eyedrops in patients with vernal keratoconjunctivitis.

DETAILED DESCRIPTION:
A total of 20 patients with bilateral symmetrical vernal keratoconjunctivitis will be included. Each patient will undergo a complete ophthalmologic evaluation. Patient will be placed at random on topical Tacrolimus 0.01% ophthalmic solution in one eye and placebo eyedrops in the fellow eye. Patients will undergo ophthalmologic examination at one week and after one month. Photos will be taken. The outcome measures include graded symptoms, graded signs, and laboratory investigations. Symptoms of itching, redness, foreign body sensation, tearing and discharge following will be recorded before and after treatment. The grading of clinical signs of conjunctival hyperemia, conjunctival papillary hypertrophy, perilimbal infiltrates, Trantas dots, superficial punctate keratopathy will be recorded before and after treatment. Conjunctival surface temperature will be determined before and after treatment. Conjunctival scrapings will be stained with Giemsa and will be assessed before and after therapy and number of eosinophils per hpf will be determined and recorded.

ELIGIBILITY:
Inclusion Criteria:

* with bilateral symmetrical palpebral and limbal vernal keratoconjunctivitis
* Patients 6-18 years of age

Exclusion Criteria:

* Pregnant patients
* Patients on systemic therapy for other allergic disorders
* Patients who cannot come for follow-up
* Patients who are on other topical medications for other comorbid ocular conditions

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The efficacy of Topical Tacrolimus in Vernal Keratoconjunctivitis | Five months
  To evaluate the efficacy of topical tacrolimus 0.01 eye drops in patients with vernal keratoconjunctivitis in symptoms of redness, itching, foreign body sensation and discharge and signs of conjunctival hyperemia,perlimbal infiltrates, Trantas dots and papillary reaction

CONTACTS AND LOCATIONS:
Overall Officials: Samir S Shoughy, Principal Investigator — THE EYE CENTER
Locations (1):
- The Eye Center, Riyadh, Saudi Arabia